CLINICAL TRIAL: NCT05731778
Title: Clinical Study to Assess Therapeutic Delay and Resolution of Induced Gingivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2018-07-IND-GING-DELAY-JG
Record Dates: First submitted 2019-07-24; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2019-04

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stannous fluoride test toothpaste (Experimental): Currently marketed as the new Colgate Total SF containing Stannous Fluoride
  Interventions: Drug: Stannous Fluoride Toothpaste
- Colgate flouride toothpaste (Placebo Comparator): Colgate Dental Cream containing Stannous Sodium Fluoride
  Interventions: Drug: Colgate fluoride toothpaste

INTERVENTIONS:
Drug: Stannous Fluoride Toothpaste — 0.454% stannous fluoride toothpaste
  Other Names: Colgate Total SF
  Arms: Stannous fluoride test toothpaste
Drug: Colgate fluoride toothpaste — 0.76 % Sodium MonoFluorophosphate (MFP)
  Other Names: Colgate Dental Cream
  Arms: Colgate flouride toothpaste

SUMMARY:
Evaluate a stannous technology for its effect on the neutrophil phenotype during an induced gingivitis state.

DETAILED DESCRIPTION:
A 9-weeks clinical study will be conducted to evaluate a stannous fluoride dentifrice for therapeutic effects that aim to delay the onset of experimental gingivitis as well as hasten the resolution of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged 18-70 years
2. In good general health, ASA I
3. No clinical signs of gingival inflammation at >90% sites observed
4. Probing Depth (PD) < 3.0 mm
5. Attachment Loss (AL) = 0 mm
6. No periodontal disease history
7. Non-smokers
8. Fluent in English

Exclusion Criteria:

1. Presence of orthodontic bands.
2. Presence of partial removal dentures.
3. Tumour(s) of the soft or the hard tissues of the oral cavity.
4. Cavitated carious lesions requiring immediate restorative treatment.
5. History of allergy to consumer or personal care products or dentifrice ingredients as determined by the dental profession monitoring the study.
6. Participation in any other clinical study or test panel with a one month period prior to entering the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-12-22 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Bleeding Index (BOP) and Oral Inflammatory Load | during patient visit over the 9 weeks
  BOP is a bleeding index standard in field, oral inflammatory load as measured by neutrophil levels in oral rinses

CONTACTS AND LOCATIONS:
Overall Officials: Michael Glogauer, DDS/PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada